CLINICAL TRIAL: NCT06098105
Title: Laparoscopic vs Ultrasound-Guided Transversus Abdominis Plane Block vs Laparoscopic Intraperitoneal Instillation of Local Anesthetic in Pediatrics Undergoing Inguinal Hernia Repair: A Randomized Controlled Trial
Brief Title: Laparoscopic vs Ultrasound-Guided Transversus Abdominis Plane Block vs Laparoscopic Intraperitoneal Instillation of Local Anesthetic in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, ِAhmed Mohamed Ibrahim, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR352/9/23
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Laparoscopic; Ultrasound; Transversus Abdominis Plane Block; Laparoscopic Intraperitoneal Instillation; Pediatrics; Inguinal Hernia Repair
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ultrasound-guided transversus abdominis plane block (Active Comparator): This group will receive Ultrasound-guided transversus abdominis plane block by using 1 ml/kg of bupivacaine 0.25% with a maximum volume of 20 mL as a control group.
  Interventions: Procedure: Ultrasound-guided transversus abdominis plane block; Drug: Bupivacaine
- Laparoscopic-assisted transversus abdominis plane block (Experimental): Patients will receive Laparoscopic-assisted transversus abdominis plane block by using 1 ml/kg of bupivacaine 0.25% with a maximum volume of 20 mL.
  Interventions: Procedure: Laparoscopic-assisted transversus abdominis plane block; Drug: Bupivacaine
- Laparoscopic-assisted intraperitoneal instillation (Experimental): This group will receive Laparoscopic-assisted intraperitoneal instillation by using 1 ml/kg of bupivacaine 0.25% with a maximum volume of 20 mL will be instilled into the peritoneal cavity immediately after gas insufflation.
  Interventions: Procedure: Laparoscopic-assisted intraperitoneal instillation; Drug: Bupivacaine

INTERVENTIONS:
Procedure: Ultrasound-guided transversus abdominis plane block — This group will receive ultrasound-guided transversus abdominis plane block by using 1 ml/kg of bupivacaine 0.25% with a maximum volume of 20 mL as a control group.
  Arms: Ultrasound-guided transversus abdominis plane block
Procedure: Laparoscopic-assisted transversus abdominis plane block — Patients will receive laparoscopic-assisted transversus abdominis plane block by using 1 ml/kg of bupivacaine 0.25% with a maximum volume of 20 mL.
  Arms: Laparoscopic-assisted transversus abdominis plane block
Procedure: Laparoscopic-assisted intraperitoneal instillation — This group will receive laparoscopic-assisted intraperitoneal instillation by using 1 ml/kg of bupivacaine 0.25% with a maximum volume of 20 mL will be instilled into the peritoneal cavity immediately after gas insufflation.
  Arms: Laparoscopic-assisted intraperitoneal instillation
Drug: Bupivacaine — bupivacaine

SUMMARY:
The aim of this study is to compare laparoscopic -assisted, ultrasound-guided transversus abdominis plane block and laparoscopic intraperitoneal instillation of local anesthetic in pediatrics undergoing inguinal hernia repair.

DETAILED DESCRIPTION:
Inguinal hernia is one of the most common pediatric surgeries. Effective and safe pain management causes fewer side effects and enables faster hospital discharge. It is also important in overcoming chronic pain in the late postoperative period.

Transversus abdominis plane block (TAPB) has emerged as a safe, simple, and inexpensive modality incorporated into many enhanced recovery pathways to achieve narcotic-sparing analgesia after bariatric surgery. TAPB was first performed through the lumbar triangle of Petit in 2001. Since that time, both ultrasound-guided (US) and laparoscopic (LAP) TAPBs have been developed to aid in proper identification of the correct plane and minimize peritoneal penetration.

ELIGIBILITY:
Inclusion Criteria:

* Age: 2 months to 7 years old
* Both sexes.
* American Society of Anesthesiologists (ASA) I-II.
* Schedule for elective unilateral inguinal hernia repair.

Exclusion Criteria:

* Patients with history of allergy.
* Hepatic and renal failure.
* Previous inguinal surgery.
* Block contraindications (e.g., infection at the site of block, bleeding disorder, or abnormalities of the sacrum).

Ages: 2 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-04-21 (Actual); Study Completion 2024-04-21 (Actual)

PRIMARY OUTCOMES:
Total postoperative pethidine consumption | 24 hours postoperatively
  The patient will be given supplementary paracetamol I.V. injection in a dose of 15 mg/kg as routine analgesia. If the FLACC score is > 3, pethidine 0.5 mg/kg.

SECONDARY OUTCOMES:
Post-operative pain scores | 24 hours postoperatively
  Face, Legs, Activity, Cry and Consolability (FLACC) scale will be used for postoperative pain assessment. This scale ranges from 0 to 10 where 0 represents no pain and 10 represents worst possible pain.
  FLACC scale will be measured at 30 minutes and then at 2, 4, 6, 12, 18 and 24 hours.
Time of first analgesia request. | 24 hours postoperatively
  Time of first analgesic requirement, which represent the time elapsed from the end of the surgery till the first request of rescue analgesia.
Incidence of adverse events | 24 hours postoperatively
  Complication related to the block or adverse events of the administered drugs.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.